CLINICAL TRIAL: NCT00006131
Title: Randomized Study of Two Doses of Oral Valacyclovir in Immunocompromised Patients With Uncomplicated Herpes Zoster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/15324; UTMB-97-120; GW-R-24; UTMB-GCRC-D085
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2007-05-24 (Estimated); Status verified 2003-12

CONDITIONS: Herpes Zoster; Immunologic Deficiency Syndromes
MeSH Terms: conditions — Herpes Zoster; Immunologic Deficiency Syndromes | interventions — Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir

SUMMARY:
OBJECTIVES:

I. Compare the efficacy and safety of two doses of oral valacyclovir in immunocompromised patients with uncomplicated herpes zoster.

II. Compare quality of life, pain, and medical resource utilization in patients treated with these 2 regimens.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, double blind study.

Patients are randomized to one of two treatment arms.

Arm I: Patients receive standard dose oral valacyclovir three times a day on Days 1-7.

Arm II: Patients receive higher dose oral valacyclovir three times a day on Days 1-7.

Both arms: Patients begin treatment within 72 hours after onset of zoster rash.

Quality of life is assessed on Days 1, 14, and 28 during study and then every 4 weeks through Week 24. Pain is assessed on Days 1-28 during study, and then weekly through Week 24. Medical resource utilization is assessed on Days 1, 8, 14, and 18 during study and then every 4 weeks through Week 24.

Patients are followed every 4 weeks through Week 24.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Patients with a clinical diagnosis of uncomplicated herpes zoster presenting within 72 hours after onset of zoster rash

No evidence of cutaneous or visceral dissemination of herpes zoster infection; cutaneous dissemination defined as at least 20 discrete lesions outside adjacent dermatomes

Must have immune dysfunction caused by any of the following: congenital immune deficiency; active malignancy of any type; collagen vascular diseases; organ or bone marrow transplantation; HIV infection; severe atopic dermatitis; received cytotoxic drugs or immunosuppressive therapy (e.g., chronic systemic corticosteroids) within past 3 months

CD4 count at least 50%

--Prior/Concurrent Therapy--

Biologic therapy: Greater than 9 months since prior bone marrow transplantation

Surgery: Greater than 9 months since prior liver or heart transplantation

Other: At least 4 weeks since prior topical or systemic anti-varicella zoster virus (anti-VZV) medications; no concurrent systemic agents with anti-VZV activity from enrollment to Day 10; no concurrent probenecid from 24 hours before the first dose of study drug until Day 10

--Patient Characteristics--

Hepatic: AST or ALT no greater than 5 times upper limit of normal

Renal: Creatinine clearance at least 30 mL/min

Other: Not pregnant or nursing; negative pregnancy test; fertile patients must use effective contraception; no history of intolerance or hypersensitivity to acyclovir, penciclovir, valacyclovir, or famciclovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 1997-01

CONTACTS AND LOCATIONS:
Overall Officials: Stephen K. Tyring, Study Chair — University of Texas
Locations (1):
- Center for Clinical Studies, Houston, Texas, United States